CLINICAL TRIAL: NCT03703336
Title: A Phase III, Randomized, Partially Double- Blind, Active Control Study to Compare the Immunogenicity and Safety of a Liquid Formulation of ROTAVIN With the Currently Licensed Frozen Formulation of the Vaccine (ROTAVIN-M1), in Healthy Vietnamese Infants
Brief Title: Phase III Study of Liquid Formulation of ROTAVIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Center for Research and Production of Vaccines and Biologicals, Vietnam (Other Government)
Collaborators: PATH (Other); National Institute of Hygiene and Epidemiology, Vietnam (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CVIA 068; VX.2018.05 (Other: Vietnam Ministry of Health)
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-11

CONDITIONS: Diarrhea; Diarrhea Rotavirus
Keywords: ROTAVIN; Rotavirus vaccine; Rotavirus; Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: Eligible infants will be randomized to receive either ROTAVIN or ROTAVIN-M1 vaccines in the ratio of 2:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROTAVIN Liquid Formulation (Experimental): Participants received two doses of ROTAVIN liquid formulation vaccine orally 8 weeks apart with the first dose administered at 60-91 days of age.
  Interventions: Biological: ROTAVIN (liquid formulation)
- ROTAVIN-M1 Frozen Formulation (Active Comparator): Participants received two doses of ROTAVIN-M1 frozen formulation vaccine orally 8 weeks apart with the first dose administered at 60-91 days of age.
  Interventions: Biological: ROTAVIN-M1 (frozen formulation)

INTERVENTIONS:
Biological: ROTAVIN (liquid formulation) — Live attenuated human rotavirus vaccine containing ≥ 2x10^6 plaque forming units (PFU) of strain G1P[8] per dose of 2 mL.
  Arms: ROTAVIN Liquid Formulation
Biological: ROTAVIN-M1 (frozen formulation) — Live attenuated human rotavirus vaccine containing ≥ 2x10^6 PFU of strain G1P[8] per dose of 2 mL.
  Arms: ROTAVIN-M1 Frozen Formulation

SUMMARY:
This study is conducted to demonstrate non-inferiority in the immunogenicity of the liquid formulation of ROTAVIN in comparison to currently licensed frozen formulation of the vaccine (ROTAVIN-M1), 28 days after the second vaccination when administered as two dose series starting at 2-3 months of age.

The study will also assess the reactogenicity of the vaccine 7 days after each vaccination and safety from first vaccination up to 4 weeks after the last vaccination.

DETAILED DESCRIPTION:
The study is designed as a phase III, randomized, partially double-blinded, active controlled study with two groups of infants receiving vaccines at the ratio of 2:1 (liquid formulation of ROTAVIN to frozen formulation ROTAVIN-M1), to compare their immunogenicity and safety. Two doses of vaccine will be administered 8 weeks apart with the first vaccine administration between 60-91 days of age. All childhood vaccines as per the Expanded Program for Immunization of the Government of Vietnam (including Diphtheria, Tetanus, Pertussis, Haemophilus influenzae type b and Hepatitis B vaccine (DTwPHib-HepB), and Oral Polio Vaccine at at 2, 3 and 4 months of age) will be allowed as per the immunization schedule.

Active surveillance for vaccine reactogenicity (solicited reactions) over the 7-day period after each vaccination, unsolicited adverse events (AEs) for 4 weeks after each vaccination and serious adverse events (SAEs) including intussusception over the period between first vaccination and four weeks after the last vaccination will be conducted for all infants.

This trial will generate immunogenicity and safety data which would be submitted to Ministry of Health in Vietnam for license of new formulation of ROTAVIN vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants as established by medical history and clinical examination before entering the study.
2. Age: 60-91 days (both days inclusive) at the time of enrollment.
3. Parental/legally acceptable representative ability and willingness to provide written informed consent.
4. Parent/legally acceptable representative who intends to remain in the area with the child during the study period.

Exclusion Criteria:

1. Presence of diarrhea or vomiting in the previous 72 hours or on the day of enrollment (temporary exclusion).
2. Presence of fever on the day of enrollment (temporary exclusion).
3. Acute disease at the time of enrollment (temporary exclusion).
4. Concurrent participation in another clinical trial at any point throughout the entire time frame for this study.
5. Presence of significant malnutrition (weight-for-height z-score < -3 SD median)
6. Presence of any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer, or autoimmune disease) as determined by medical history and / or physical examination which would compromise the participant's health or is likely to result in nonconformance to the protocol.
7. History of congenital abdominal disorders, intussusception, or abdominal surgery.
8. Known or suspected impairment of immunological function based on medical history and physical examination.
9. Household contact with an immunosuppressed individual or pregnant woman.
10. Prior receipt of rotavirus or an intent to receive this vaccine from outside of the study center during study participation.
11. Prior receipt of Expanded Program on Immunization (EPI) vaccination during past 7 days or plan to receive them within next 7 days.
12. A known sensitivity or allergy to any components of the study vaccine.
13. History of allergy to antibiotic kanamycin.
14. Clinically detectable significant congenital or genetic defect.
15. History of persistent diarrhea (defined as diarrhea that lasts 14 days or longer).
16. Receipt of immunoglobulin therapy and / or blood products since birth or planned administration during the study period.
17. History of chronic administration (defined as more than 14 days) of immunosuppressants including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study.
18. Any medical condition in the parent/legally acceptable representative or infant which, in the judgment of the Investigator, would interfere with or serves as a contraindication to protocol adherence.

Ages: 60 Days to 91 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 825 (Actual)
Dates: Start 2019-03-16 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Rathi, MD, Study Director — PATH India
Locations (2):
- Vietnam (2):
  - CDC Nam Dinh, Nam Định
  - CDC Quang Ninh, Quang Ninh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thiem VD, Anh DD, Ha VH, Hien ND, Huong NT, Nga NT, Thang TC, McNeal MM, Meyer N, Pham HL, Huong NM, Gompana G, Cassels F, Tang Y, Flores J, Rathi N. Safety and immunogenicity of two formulations of rotavirus vaccine in Vietnamese infants. Vaccine. 2021 Jul 22;39(32):4463-4470. doi: 10.1016/j.vaccine.2021.06.056. Epub 2021 Jul 1. PMID 34218961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by the National Institute of Hygiene and Epidemiology (NIHE) at 12 health centers in one district in the Nam Dinh province and at 12 health centers in one district in the Quang Ninh province in Vietnam.
Pre-assignment Details: Infants were allocated to one of the two groups at a ratio of 2:1 to receive either the ROTAVIN liquid formulation or the frozen formulation ROTAVIN-M1.
Period: Overall Study
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
Started | 552 | 273
Received Dose 1 | 552 | 273
Received Dose 2 | 518 | 263
Safety Population (The safety population was defined as all participants in the enrolled population who received a study vaccination. One participant was randomized to ROTAVIN but instead received ROTAVIN-M1 and was therefore analyzed in ROTAVIN-M1 group for safety population based on the actual treatment received.) | 551 | 274
Completed | 514 | 259
Not Completed | 38 | 14
Not completed — Parent withdrew consent | 29 | 8
Not completed — Migration | 3 | 3
Not completed — Protocol Violation | 3 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population, as treated
Groups:
- Total: Total of all reporting groups
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation | Total
Number analyzed (Participants) | 551 | 274 | 825
Age, Continuous [Mean (Standard Deviation); unit: days] | 74.7 (8.63) | 75.2 (9.15) | 74.8 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 144 | 420
  Male | 275 | 130 | 405
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Vietnamese | 551 | 274 | 825
Province [Count of Participants; unit: Participants]
  Nam Dinh province | 251 | 124 | 375
  Quang Ninh province | 300 | 150 | 450

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration (GMC) of Serum Anti-rotavirus Immunoglobulin A (IgA) Antibodies 28 Days After Second Vaccination
Description: Serum anti-rotavirus IgA antibodies were measured using a validated enzyme linked immunosorbent assay (ELISA) at the Cincinnati Children's Hospital Medical Center (CCHMC), Division of Infectious Diseases in Cincinnati, Ohio USA.
Time Frame: Day 85 (28 days after the second vaccination)
Population: Immunogenicity assays were conducted on the subset of participants enrolled at Quang Ninh.
  The Per-Protocol (PP) population was defined as randomized participants who received a study vaccination, provided at least one evaluable serum sample, and who correctly received study vaccine per randomization with no major protocol deviations that were determined to potentially interfere with the immunogenicity assessment of the study vaccines.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
Number analyzed (Participants) | 267 | 135
U/mL | 48.25 [40.59 to 57.37] | 35.04 [27.34 to 44.91]
Statistical Analysis 1: Comparison: ROTAVIN Liquid Formulation vs ROTAVIN-M1 Frozen Formulation; Test type: Non-Inferiority — If the lower limit of the 95% confidence interval (CI) of the ratio of GMCs between the ROTAVIN and ROTAVIN-M1 groups were to be larger than 1/2, ROTAVIN was considered to be non-inferior to the licensed frozen formulation of the vaccine (ROTAVIN-M1); GMC Ratio = 1.38, 95% CI 2-sided [1.02 to 1.86] — Log10-transformed IgA concentrations were used to construct a 2-sided 95% CI for the mean difference between the arms using t-distribution. The mean difference and 95% CI were exponentiated to obtain the GMC ratio and corresponding 95% CI

2. Primary Outcome: Number of Participants With Solicited Reactions Within 7 Days of Vaccination
Description: Solicited post-vaccination reactogenicity included fever, diarrhea, vomiting, decreased appetite, irritability, and decreased activity level during the seven-day period after each vaccination. Parents were asked to record reactions on a post-immunization diary card.
  Solicited reactions were graded for severity on a scale from mild to severe based on the level of symptoms.
Time Frame: 7 days after each vaccination (Days 1 to 8 and 57 to 64)
Population: Safety population, as treated
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
Number analyzed (Participants) | 551 | 274
Participants
  Any solicited reaction | 195 | 102
  Fever | 37 | 23
  Diarrhoea | 57 | 27
  Vomiting | 78 | 33
  Decreased appetite | 68 | 28
  Irritability | 92 | 48
  Decreased activity level | 35 | 23
  Mild severity | 173 | 85
  Moderate severity | 61 | 37
  Severe severity | 22 | 8

3. Secondary Outcome: Percentage of Participants With Seroconversion 28 Days After the Second Vaccination
Description: Seroconversion is defined as a post-vaccination serum anti-rotavirus IgA antibody concentration of at least 20 U/mL if the baseline concentration was < 20 U/mL or a post- vaccination serum anti-rotavirus IgA antibody concentration of ≥ 4-fold baseline level if the baseline concentration was ≥ 20 U/mL.
Time Frame: 28 days after the second vaccination (Day 85)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
Number analyzed (Participants) | 267 | 135
percentage of participants | 70.4 [64.54 to 75.82] | 64.4 [55.75 to 72.49]
Statistical Analysis 1: Comparison: ROTAVIN Liquid Formulation vs ROTAVIN-M1 Frozen Formulation; Test type: Other; Percentage Difference = 6.0, 95% CI 2-sided [-3.57 to 15.87]

4. Secondary Outcome: Percentage of Participants With Seropositivity at Baseline and 28 Days After the Second Vaccination
Description: Seropositivity is defined as serum IgA antibody concentration ≥ 20 U/mL
Time Frame: Baseline (Day 1) and at 28 days after the second vaccination (Day 85)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
Number analyzed (Participants) | 267 | 135
percentage of participants
  Day 1 | 0.4 [0.01 to 2.07] | 0.0 [0.00 to 2.70]
  Day 85 | 70.8 [64.93 to 76.17] | 64.4 [55.75 to 72.49]
Statistical Analysis 1: Comparison: ROTAVIN Liquid Formulation vs ROTAVIN-M1 Frozen Formulation; Percentage Difference on Day 1; Test type: Other; Percentage Difference = 0.4, 95% CI 2-sided [-2.40 to 2.09]
Statistical Analysis 2: Comparison: ROTAVIN Liquid Formulation vs ROTAVIN-M1 Frozen Formulation; Percentage Difference on Day 85; Test type: Other; Percentage Difference = 6.3, 95% CI 2-sided [-3.19 to 16.23]

5. Secondary Outcome: Number of Participants With Immediate Adverse Events (AEs)
Description: After each vaccination participants were observed at the clinic site for at least 30 minutes to check for any immediate AEs including episodes of vomiting and allergic reaction to vaccine. Immediate AEs include all reactions that occurred within 30 minutes of each vaccination.
  Reactions were graded for severity per the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, version 2.1, of the US National Institute of Health:
  Grade 1: Mild symptoms causing no or minimal interference with usual social & functional activities; intervention not indicated.
  Grade 2: Moderate symptoms causing greater than minimal interference with usual activities; intervention indicated.
  Grade 3: Severe symptoms causing inability to perform usual activities; intervention or hospitalization indicated.
  Grade 4: Potentially life-threatening symptoms; intervention indicated to prevent permanent impairment, persistent disability, or death
  Grade 5: Death
Time Frame: Within 30 minutes after each vaccination on Day 1 and Day 57
Population: Safety population, as treated
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
Number analyzed (Participants) | 551 | 274
Participants
  Any immediate adverse event | 2 | 0
  Immediate AEs occurring after dose 1 | 0 | 0
  Immediate AEs occurring after dose 2 | 2 | 0
  Vomiting | 1 | 0
  Pyrexia | 1 | 0
  Mild Immediate AEs | 2 | 0
  Moderate Immediate AEs | 0 | 0
  Severe Immediate AEs | 0 | 0
  Life-threatening Immediate AEs | 0 | 0
  Death | 0 | 0

6. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An unsolicited AE was any AE that occurred after vaccination, whether or not deemed "related" to the product, that was not solicited, or, any solicited reaction that started after 7 days post-vaccination. Severity of unsolicited AEs was graded per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, version 2.1.
  Grade 1: Mild symptoms causing no or minimal interference with usual social & functional activities; intervention not indicated
  Grade 2: Moderate symptoms causing greater than minimal interference with usual activities; intervention indicated
  Grade 3: Severe symptoms causing inability to perform usual activities; intervention or hospitalization indicated
  Grade 4: Potentially life-threatening symptoms; intervention indicated to prevent permanent impairment, persistent disability, or death
  Grade 5: Death
  The clinician classified the causality of each AE as related if there was reasonable possibility that the product caused the event.
Time Frame: From vaccination through 28 days after each dose (Days 1 to 28 and 57 to 85)
Population: Safety population, as treated
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
Number analyzed (Participants) | 551 | 274
Participants
  Any unsolicited adverse events | 292 | 154
  Mild adverse events | 191 | 103
  Moderate adverse events | 132 | 63
  Severe adverse events | 20 | 10
  Life-threatening adverse events | 0 | 0
  Death | 0 | 0
  Related to study vaccine | 2 | 0
  Unrelated to study vaccine | 291 | 154

7. Secondary Outcome: Number of Participants With Serious Adverse Events Including Intussusception
Description: All Serious adverse events (SAEs), including cases of intussusception, were recorded at all time points between first vaccination and last visit. An SAE was defined as any untoward medical occurrence that:
  * Resulted in death,
  * Was life threatening,
  * Required inpatient hospitalization or prolongation of existing hospitalization,
  * Resulted in persistent or significant disability / incapacity,
  * Was a congenital anomaly or a birth defect,
  * Medically important event
  Investigator-confirmed cases of intussusception also qualified as an SAE in this study. Intussusception is the infolding (telescoping) of one segment of the intestine within another, usually resulting in a blockage of the intestine.
Time Frame: From first vaccination through 28 days after the last vaccination; 85 days
Population: Safety population, as treated
Measure: Count of Participants; unit: Participants
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
Number analyzed (Participants) | 551 | 274
Participants
  Any serious adverse event | 23 | 14
  SAEs related to study vaccine | 3 | 3
  SAEs unrelated to study vaccine | 20 | 11
  Intussusception | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events and mortality are reported from the first vaccination date until 28 days after last dose; 85 days. Other adverse events are reported up to 28 days after each dose (Days 1-28 and 57 to 85)
Description: Safety population, as treated One participant was randomized to ROTAVIN but instead received ROTAVIN-M1 and was therefore analyzed in the ROTAVIN-M1 group for safety based on the actual treatment received.
Arm/Group | ROTAVIN Liquid Formulation | ROTAVIN-M1 Frozen Formulation
All-Cause Mortality (participants affected / at risk) | 0/551 | 0/274
Serious Adverse Events (participants affected / at risk) | 23/551 | 14/274
Other Adverse Events (participants affected / at risk) | 292/551 | 154/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ROTAVIN Liquid Formulation (N=551) | ROTAVIN-M1 Frozen Formulation (N=274)
Pneumonia (Infections and infestations) | 8 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Bronchiolitis (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Pertussis (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 3 | 5
Enteritis (Gastrointestinal disorders) | 1 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diarrhoea infectious (Gastrointestinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ROTAVIN Liquid Formulation (N=551) | ROTAVIN-M1 Frozen Formulation (N=274)
Pyrexia (General disorders) | 226 | 112
Vaccination site inflammation (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 22 | 7
Nasopharyngitis (Infections and infestations) | 12 | 10
Bronchitis (Infections and infestations) | 13 | 7
Pneumonia (Infections and infestations) | 8 | 4
Pharyngitis (Infections and infestations) | 4 | 2
Otitis media (Infections and infestations) | 2 | 2
Rhinitis (Infections and infestations) | 3 | 1
Bronchiolitis (Infections and infestations) | 3 | 0
Oral candidiasis (Infections and infestations) | 2 | 1
Otitis media acute (Infections and infestations) | 2 | 1
Conjunctivitis (Infections and infestations) | 1 | 1
Furuncle (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lymph node tuberculosis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 1 | 0
Roseola (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 6
Dyspepsia (Gastrointestinal disorders) | 11 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Diarrhoea infectious (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal infection (Gastrointestinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 2 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Nasal cavity packing (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03703336/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT03703336/SAP_001.pdf